CLINICAL TRIAL: NCT05922579
Title: Treatment Preferences for Somatuline® Injector Devices: A Discrete Choice Experiment (DCE) of Patients With Neuroendocrine Tumors (NETs) and Nurses in the United States (US) and Canada
Brief Title: A Study to Collect the Somatuline® Injector Device Preferences of Patients Living With Neuroendocrine Tumor (NET) and Nurses Involved in the Care of Patients With NET
Status: Terminated | Type: Observational
Why Stopped: Significant and complex challenges had since been identified during recent testing phases. After their assessment, Ipsendecided to discontinue development of this motorized device in order to not burden participants.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-52030-458
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the treatment preferences of patients with Neuroendocrine Tumors (NETS) and nurses who are involved in the care of individuals with NETs. NETs are a type of abnormal growth that can develop in various parts of the body, such as the lungs, pancreas, gastrointestinal tract, or other organs.

NETs originate from specialized cells called neuroendocrine cells, which are responsible for producing hormones in our bodies.

The study focuses on hypothetical preferences regarding the use of two different type of devices for administering Somatostatin analogues (SSAs), which could be used in the treatment of NETs.

SSAs work by imitating the actions of a hormone called somatostatin that naturally exists in our bodies. These treatment help to control the symptoms of NETs by blocking the release of hormones from the tumor cells.

The devices under consideration are a motorized injector versus a manual injector.

Participants in the study will be asked to take part in:

1. An interview based on a draft survey: 60-minute interview over videocall, to examine participants understanding of the online survey; or
2. Final online survey: 30-minute online survey. This involves presenting patients and nurses with different treatment options and asking them to choose their preferred option.

By analysing the choices made by participants, researchers can understand which attributes of the injector devices are most important to patients and nurses.

Individual participation is limited to the interview based on a draft survey (60 minutes) or the final online survey (30 minutes).

No further participation is required beyond this.

ELIGIBILITY:
Inclusion Criteria:

Patients (cognitive interviews)

* Aged 18 years or over
* Reside in the US or Canada
* Have been diagnosed with NETs by a healthcare professional (based on self-report and confirmed via data quality checks)
* Have any SSA treatment experience in the past 2 years
* Be fluent in spoken and written English
* Have read, understood, and consented to participate in the study
* Be able to complete the survey on a standard-sized tablet device (minimum 10 inches), laptop, or desktop computer
* Be able and willing to screenshare with the interviewer

Patients (online survey and DCE)

* Aged 18 years or over
* Reside in the US or Canada
* Have been diagnosed with NETs by a healthcare professional (based on self-report and confirmed via data quality checks)
* Have any SSA treatment experience in the past 2 years
* Be fluent in spoken and written English
* Have read, understood, and consented to participate in the study
* Be able to complete the survey on a standard-sized tablet device (minimum 10 inches), laptop, or desktop computer
* Have not participated in the cognitive interviews

Nurses (cognitive interviews)

* Reside in the US or Canada
* Nurse with at least 12 months experience caring for patients with NETs
* Have administered at least one long-acting SSA injection to a patient with NETs in the past 12 months
* Be fluent in spoken and written English
* Have read, understood, and consented to participate in the study
* Be able to complete the survey on a standard-sized tablet device (minimum 10 inches), laptop, or desktop computer
* Be able and willing to screenshare with the interviewer

Nurses (online survey and DCE)

* Reside in the US or Canada
* Nurse with at least 12 months experience caring for patients with NETs
* Have administered at least one long-acting SSA injection to a patient with NETs in the past 12 months
* Be fluent in spoken and written English or Canadian French
* Have read, understood, and consented to participate in the study
* Be able to complete the survey on a standard-sized tablet device (minimum 10 inches), laptop, or desktop computer
* Have not participated in the cognitive interviews

Exclusion Criteria:

* No access to internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes:
  1. patients with NETs in the US or Canada having had any SSA treatment experience in the past 2 years
  2. nurses who treat NETs in the US or Canada, having administered at least one long-acting SSA injection to a patient with NETs in the past 12 months
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Attribute importance | At the end of the survey completion (approximatively 3 months)
  Using the data from the survey scenarios (the DCE component of the survey) the DCE model estimates the parameters (β's) for each feature (attribute) level. These β's describe the magnitude and direction of influence of each of the attribute (levels) in the choice context. The β's can include negative and positive values which indicate the direction of the effect in relation to the attribute levels.
Relative attribute importance | At the end of the survey completion (approximatively 3 months)
  Attribute importance is described by the magnitude of the β's (i.e., the size of the values). The magnitude of the β's are interpreted and understood relative to each other (relative attribute importance).

SECONDARY OUTCOMES:
Measures of segmentation | At the end of the survey completion (approximatively 3 months)
  Identify which patients (e.g., age, gender, tumor grade, carcinoid syndrome status, treatment history) and nurses characteristics (e.g., years of experience, caseload, public or private place of work, NETs specialist clinic or not) are predictive of the assessment of the benefits and risks of treatment options (segmentation)
  Segmentation: The econometric methods to be employed will recognise that preferences may vary across participants, even after controlling for observed characteristics like treatment experiences. This allows for preference heterogeneity (i.e., different participants can have different marginal utility or parameter weights for each of the features).
Predicted uptake (preference share) | At the end of the survey completion (approximatively 3 months)
  Preference share: Predicted uptake for the different treatments available will be calculated, based on attribute importance..

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- CAPPRE, Sydney, Australia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/